CLINICAL TRIAL: NCT01906047
Title: Impact of Chronic Air Pollution on Non-cystic Fibrosis Bronchiectasis
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Dr. Lieven Dupont, Prof. Dr. Lieven Dupont, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: NCFB chronic pollution
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Bronchiectasis
Keywords: Non-cystic fibrosis bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
We aim at investigation the impact of chronic air pollution exposure on non-cystic fibrosis bronchiectasis outcome.

DETAILED DESCRIPTION:
* Patient files will be search for time of death and cause of death.
* Other variables will be collected: bacterial culture results, therapy, gender, age, etc.
* These data will be linked with pollution data: trafic load, distance to major road, etc.

ELIGIBILITY:
Inclusion Criteria:

* HRCT diagnosis of bronchiectasis
* recurrent infections or chronic sputum production
* patients between 18 and 65 years old.

Exclusion Criteria:

* Cystic Fibrosis
* Tumoral disease
* Traction bronchiectasis due to interstitial lung disease
* patients older than 65 years or younger than 18 years at recruitment
* COPD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a HRCT diagnosis of bronchiectasis and do not have a diagnosis of cystic fibrosis. They also need to have typical bronchiectatic disease (recurrent infections and sputum).
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2006-06; Primary Completion 2012-10 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Death | 6 years
  From June 2006 till October 2012, enrolled patients' medical file will be screened if death has occurred. If so, cause of death will be search for in the patients' file.

CONTACTS AND LOCATIONS:
Overall Officials: Lieven J Dupont, MD, PhD, Principal Investigator — UZ Leuven; Pieter C Goeminne, MD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] Goeminne PC, Bijnens E, Nemery B, Nawrot TS, Dupont LJ. Impact of traffic related air pollution indicators on non-cystic fibrosis bronchiectasis mortality: a cohort analysis. Respir Res. 2014 Sep 3;15(1):108. doi: 10.1186/s12931-014-0108-z. PMID 25183428